CLINICAL TRIAL: NCT04841863
Title: Secondary Prevention of Dug-related Problems Through Patient Empowerment Through Digital Health
Brief Title: Secondary Prevention of Dug-related Problems Through Digital Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Ana Juanes, Doctor, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIBSP-COD-2019-46
Record Dates: First submitted 2021-03-18; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Drug-Related Problems
Keywords: DRP; Digital Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug Code Active Patient o DCAP (Active Comparator): Inclusion in the active group involves the use of MyPlan digital health tool that aims to improve clinical-patient communication, enahnce patient empowerment, improve early detection of side effects and allows professionals to individualize interventions.
  Patients will receive follow-up by videoconference 48 hours after discharge and in the phase II, at 6 and 12 months after discharge.
  Interventions: Device: MyPlan digital health platform
- Standard care (Placebo Comparator): Inclusion in the control group do not involves the use of MyPlan digital health tool. Patients will receive the standard of care.
  Patients will receive follow-up by videoconference 48 hours after discharge and in the phase II, at 6 and 12 months after discharge.
  Interventions: Other: Satndard care

INTERVENTIONS:
Device: MyPlan digital health platform — Inclusion in the active group involves the use of MyPlan digital health tool that aims to improve clinical-patient communication, enahnce patient empowerment, improve early detection of side effects and allows professionals to individualize interventions.
  Arms: Drug Code Active Patient o DCAP
Other: Satndard care — Inclusion in the control group do not involves the use of MyPlan digital health tool. Patients will receive the standard of care.
  Arms: Standard care

SUMMARY:
The purpose of this study is to evaluate the clinical impact of a program for the secondary prevention of drug-realted problems (DRP) focused on the patient empowerment through Digital Health in patients who visit the Emergency Department (ED) of the Hospital de la Santa Creu i Sant Pau (HSCiSP) for a health problem related to medication in terms of readmissions, revisits and quality of life.

DETAILED DESCRIPTION:
After being infomed about the estudy and potential risks, all patients who meet the eligibility requirements and giving written informed consent, will be randomized.

The project is structured in two consecutive phases.

1. st Phase: 3-month randomized pilot study. Patients will be randomized with a 1:1 distribution to be included in the Drug Code Active Patient or DCAP (intervention group) or to receive usual care (control group). The pilot study will confirm whether the proposed methodology is feasible to implement it on a large scale, as well as providing the information necessary to calculate the sample of patients according to the main objective of the study.
2. nd Phase: Randomized clinical trial lasting 18 months (6 of which will be recruitment and 12 months follow-up) following the methodology described for the pilot in a larger sample of patients until the calculated sample size is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Visit ED for a DRP caused bu a drug of the ATC groups A, B, C or N.
* Be independent for activities of daily living (equivalent to Barthel 100).
* Have a Chalson Comorbidity Index 2 <= 3.
* Not present cognitive impairment.
* Be directly responsible for pharmacotherapy.
* Have a mobile device compatible with the MyPlan mobile application and access to Wi-Fi or mobile data, enabling the use of the technology platform from home.

Exclusion Criteria:

* Important language barrier.
* Impossibility of carrying out the necessary questionnaires or interviews defined in the methods of this study.
* Mental pathology that makes the autonomous use of technology impossible or that represents a safety problem for the patient according to clinical criteria.
* Patients not residing in the territory who cannot be followed-up later.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Clinical impact of a digitial health tool for secondary prevention of DRP focused on patient empowerment. | Baseline, 48h after discharge, 30-day and 90-day after discharge (in phase I, Pilot Trial)
  Change in clinical impact during the follow-up time will be evaluated in terms of number of readmissions, number of revisits and quality of life (based on the result obtained in the EQ-5D-3L51 questionnaire)
Clinical impact of a digitial health tool for secondary prevention of DRP focused on patient empowerment. | Baseline, 48h after discharge, 6-month and 12-month after discharge (in phase II, Clinical Trial)
  Change in clinical impact during the follow-up time will be evaluated in terms of number of readmissions, number of revisits and quality of life (based on the result obtained in the EQ-5D-3L51 questionnaire)

SECONDARY OUTCOMES:
Identify, classify, and quantify DRP that cause urgent care in a tertiary hospital in this patient population. | Baseline
  Type of DRP that promotes ED visits characterized according to the three dimensions of the Third Consensus of Granada (Need, Effectiveness and Safety)
Identify risk factors for ED visits related to DRP | Baseline
  Age, sex, social and familiar environment, blood presure (mmHg), heart frequency (bpm), Hb1Ac (%), pain (visual analog scale), weight (kg) and height (cm), chronic kidney disease, number of drugs at admission and at discharge, number of chronic health problems.
Identify which groups of drugs are more frequently associated to DRP | Baseline
  Using ATC group classification
Change in the patient therapeutic adherence | Baseline, 48h after discharge, 30-day and 90-day after discharge (in phase I, Pilot Trial)
  Active days on the MyPlan platform, functionalities used, number of queries made through platform messaging
Change in the patient therapeutic adherence | Baseline, 48h after discharge, 6-month and 12-month after discharge (in phase II, Clinical Trial)
  Active days on the MyPlan platform, functionalities used, number of queries made through platform messaging
Mesure therapeutic complexity | Baseline
  Using patient Medication Regimen Complexity Index (pMRCI-S) questionnaire
Identify predictive factors of a greater capacity for digital empowerment. | Baseline
  Using the CAMBADOS questionnaire
Measure the usability and satisfaction of patients, caregivers and professionals of the MyPlan digital health tool | 90-day after discharge (in phase I, Pilot Trial)
  Using the TrilemaSalud questionnaire
Measure the usability and satisfaction of patients, caregivers and professionals of the MyPlan digital health tool | 12-month after discharge (in phase II, Clinical Trial)
  Using the TrilemaSalud questionnaire
Change in the quality of life of patients in the active group | Baseline, 30-day and 90-day after discharge (in phase I, Pilot Trial)
  Using the EQ-5D-3L51 questionnaire
Change in the quality of life of patients in the active group | Baseline, 6-month and 12-month after discharge (in phase II, Clinical Trial)
  Using the EQ-5D-3L51 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Laia López Vinardell, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Monitor clinical trial will have access to all study data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be avaliable for monitor during the whole study period
Access Criteria: All data may be analysed and revised during the whole study period by the monitor and investigators

REFERENCES:
- [Background] Lazarou J, Pomeranz BH, Corey PN. Incidence of adverse drug reactions in hospitalized patients: a meta-analysis of prospective studies. JAMA. 1998 Apr 15;279(15):1200-5. doi: 10.1001/jama.279.15.1200. PMID 9555760
- [Background] Patel P, Zed PJ. Drug-related visits to the emergency department: how big is the problem? Pharmacotherapy. 2002 Jul;22(7):915-23. doi: 10.1592/phco.22.11.915.33630. PMID 12126224
- [Background] Baena MI, Fajardo PC, Pintor-Marmol A, Faus MJ, Marin R, Zarzuelo A, Martinez-Olmos J, Martinez-Martinez F. Negative clinical outcomes of medication resulting in emergency department visits. Eur J Clin Pharmacol. 2014 Jan;70(1):79-87. doi: 10.1007/s00228-013-1562-0. Epub 2013 Oct 3. PMID 24091839
- [Background] Castro I, Guardiola JM, Tuneu L, Sala ML, Faus MJ, Mangues MA. Drug-related visits to the emergency department in a Spanish university hospital. Int J Clin Pharm. 2013 Oct;35(5):727-35. doi: 10.1007/s11096-013-9795-7. Epub 2013 May 22. PMID 23695594
- [Background] Banerjee J, Conroy S, Cooke MW. Quality care for older people with urgent and emergency care needs in UK emergency departments. Emerg Med J. 2013 Sep;30(9):699-700. doi: 10.1136/emermed-2012-202080. Epub 2012 Dec 18. No abstract available. PMID 23250895
- [Background] Hamilton HJ, Gallagher PF, O'Mahony D. Inappropriate prescribing and adverse drug events in older people. BMC Geriatr. 2009 Jan 28;9:5. doi: 10.1186/1471-2318-9-5. PMID 19175914
- [Background] Leendertse AJ, Egberts AC, Stoker LJ, van den Bemt PM; HARM Study Group. Frequency of and risk factors for preventable medication-related hospital admissions in the Netherlands. Arch Intern Med. 2008 Sep 22;168(17):1890-6. doi: 10.1001/archinternmed.2008.3. PMID 18809816
- [Background] Gheewala PA, Peterson GM, Curtain CM, Nishtala PS, Hannan PJ, Castelino RL. Impact of the pharmacist medication review services on drug-related problems and potentially inappropriate prescribing of renally cleared medications in residents of aged care facilities. Drugs Aging. 2014 Nov;31(11):825-35. doi: 10.1007/s40266-014-0208-y. PMID 25187228
- [Background] Patterson SM, Cadogan CA, Kerse N, Cardwell CR, Bradley MC, Ryan C, Hughes C. Interventions to improve the appropriate use of polypharmacy for older people. Cochrane Database Syst Rev. 2014 Oct 7;(10):CD008165. doi: 10.1002/14651858.CD008165.pub3. PMID 25288041
- [Background] Campins L, Serra-Prat M, Palomera E, Bolibar I, Martinez MA, Gallo P. Reduction of pharmaceutical expenditure by a drug appropriateness intervention in polymedicated elderly subjects in Catalonia (Spain). Gac Sanit. 2019 Mar-Apr;33(2):106-111. doi: 10.1016/j.gaceta.2017.09.002. Epub 2017 Nov 20. PMID 29162290
- [Background] Perez Menendez-Conde C, Bermejo Vicedo T, Delgado Silveira E, Carretero Accame E. Adverse drug reactions which provoke hospital admission. Farm Hosp. 2011 Sep-Oct;35(5):236-43. doi: 10.1016/j.farma.2010.08.003. Epub 2011 May 12. English, Spanish. PMID 21570331
- [Background] Donaldson LJ, Kelley ET, Dhingra-Kumar N, Kieny MP, Sheikh A. Medication Without Harm: WHO's Third Global Patient Safety Challenge. Lancet. 2017 Apr 29;389(10080):1680-1681. doi: 10.1016/S0140-6736(17)31047-4. No abstract available. PMID 28463129
- [Background] Lancaster K, Abuzour A, Khaira M, Mathers A, Chan A, Bui V, Lok A, Thabane L, Dolovich L. The Use and Effects of Electronic Health Tools for Patient Self-Monitoring and Reporting of Outcomes Following Medication Use: Systematic Review. J Med Internet Res. 2018 Dec 18;20(12):e294. doi: 10.2196/jmir.9284. PMID 30563822
- [Background] Martinez-Pillado M, Said-Criado I, Regueiro-Martinez A, Rodriguez IC. E-young chronics y e-senior chronics como nuevos modelos para la atencion a la cronicidad. J Healthc Qual Res. 2018 May-Jun;33(3):119-120. doi: 10.1016/j.jhqr.2018.07.001. No abstract available. Spanish. PMID 30328812
- [Background] Park LG, Howie-Esquivel J, Dracup K. A quantitative systematic review of the efficacy of mobile phone interventions to improve medication adherence. J Adv Nurs. 2014 Sep;70(9):1932-1953. doi: 10.1111/jan.12400. Epub 2014 Apr 1. PMID 24689978
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Ritterband LM, Andersson G, Christensen HM, Carlbring P, Cuijpers P. Directions for the International Society for Research on Internet Interventions (ISRII). J Med Internet Res. 2006 Sep 29;8(3):e23. doi: 10.2196/jmir.8.3.e23. PMID 17032639
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Piette JD, Striplin D, Marinec N, Chen J, Trivedi RB, Aron DC, Fisher L, Aikens JE. A Mobile Health Intervention Supporting Heart Failure Patients and Their Informal Caregivers: A Randomized Comparative Effectiveness Trial. J Med Internet Res. 2015 Jun 10;17(6):e142. doi: 10.2196/jmir.4550. PMID 26063161
- [Background] Piette JD, List J, Rana GK, Townsend W, Striplin D, Heisler M. Mobile Health Devices as Tools for Worldwide Cardiovascular Risk Reduction and Disease Management. Circulation. 2015 Nov 24;132(21):2012-27. doi: 10.1161/CIRCULATIONAHA.114.008723. PMID 26596977
- [Background] Comin-Colet J, Enjuanes C, Verdu-Rotellar JM, Linas A, Ruiz-Rodriguez P, Gonzalez-Robledo G, Farre N, Moliner-Borja P, Ruiz-Bustillo S, Bruguera J. Impact on clinical events and healthcare costs of adding telemedicine to multidisciplinary disease management programmes for heart failure: Results of a randomized controlled trial. J Telemed Telecare. 2016 Jul;22(5):282-95. doi: 10.1177/1357633X15600583. Epub 2015 Sep 7. PMID 26350543
- [Background] de la Torre-Diez I, Lopez-Coronado M, Vaca C, Aguado JS, de Castro C. Cost-utility and cost-effectiveness studies of telemedicine, electronic, and mobile health systems in the literature: a systematic review. Telemed J E Health. 2015 Feb;21(2):81-5. doi: 10.1089/tmj.2014.0053. Epub 2014 Dec 4. PMID 25474190
- [Background] Wei L, Yang X, Li J, Liu L, Luo H, Zheng Z, Wei Y. Effect of pharmaceutical care on medication adherence and hospital admission in patients with chronic obstructive pulmonary disease (COPD): a randomized controlled study. J Thorac Dis. 2014 Jun;6(6):656-62. doi: 10.3978/j.issn.2072-1439.2014.06.20. PMID 24976987
- [Background] Koshman SL, Charrois TL, Simpson SH, McAlister FA, Tsuyuki RT. Pharmacist care of patients with heart failure: a systematic review of randomized trials. Arch Intern Med. 2008 Apr 14;168(7):687-94. doi: 10.1001/archinte.168.7.687. PMID 18413550
- [Background] Ravn-Nielsen LV, Duckert ML, Lund ML, Henriksen JP, Nielsen ML, Eriksen CS, Buck TC, Pottegard A, Hansen MR, Hallas J. Effect of an In-Hospital Multifaceted Clinical Pharmacist Intervention on the Risk of Readmission: A Randomized Clinical Trial. JAMA Intern Med. 2018 Mar 1;178(3):375-382. doi: 10.1001/jamainternmed.2017.8274. PMID 29379953
- [Background] Gomis-Pastor M, Roig Mingell E, Mirabet Perez S, Brossa Loidi V, Lopez Lopez L, Diaz Bassons A, Aretio Pousa A, Feliu Ribera A, Ferrero-Gregori A, Guirado Perich L, Mangues Bafalluy MA. Multimorbidity and medication complexity: New challenges in heart transplantation. Clin Transplant. 2019 Oct;33(10):e13682. doi: 10.1111/ctr.13682. Epub 2019 Aug 28. PMID 31368585
- [Background] Anglada-Martinez H, Martin-Conde M, Rovira-Illamola M, Sotoca-Momblona JM, Sequeira E, Aragunde V, Moreno MA, Catalan M, Codina-Jane C. Feasibility and Preliminary Outcomes of a Web and Smartphone-Based Medication Self-Management Platform for Chronically Ill Patients. J Med Syst. 2016 Apr;40(4):99. doi: 10.1007/s10916-016-0456-y. Epub 2016 Feb 12. PMID 26872781
- [Background] Tickle-Degnen L. Nuts and bolts of conducting feasibility studies. Am J Occup Ther. 2013 Mar-Apr;67(2):171-6. doi: 10.5014/ajot.2013.006270. PMID 23433271
- [Background] Eysenbach G; CONSORT-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of Web-based and mobile health interventions. J Med Internet Res. 2011 Dec 31;13(4):e126. doi: 10.2196/jmir.1923. PMID 22209829
- [Background] Chen CE, Harrington RA, Desai SA, Mahaffey KW, Turakhia MP. Characteristics of Digital Health Studies Registered in ClinicalTrials.gov. JAMA Intern Med. 2019 Jun 1;179(6):838-840. doi: 10.1001/jamainternmed.2018.7235. PMID 30801617